CLINICAL TRIAL: NCT05590364
Title: Interventional, Post-marketing, Local, Mono-centric Study for Evaluation of Aesthetic Performance and Tolerance of an Injective Intradermal Treatment for the Skin Roughness and Laxity of Back of the Hands
Brief Title: Aesthetic Performance and Tolerance of an Injective Intradermal Treatment for the Skin Roughness and Laxity of Back of the Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IBSA Farmaceutici Italia Srl (Industry)
Collaborators: Derming SRL (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E0122
Record Dates: First submitted 2022-09-27; First posted 2022-10-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-11

CONDITIONS: Skin Laxity; Skin Roughness
Keywords: Skin laxity; Skin roughness; Profhilo Body; Hyaluronic Acid; Hybrid Cooperative Complexes
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: 55 subjects undergoing Profhilo Body treatment in the back of the hands, 3 visits: Day 0 (treatment) Day 30 (1 month after Day 0 treatment) Day 120 (4 months after Day 0 - follow-up).
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Profhilo® Body treatment group (Experimental): 1.5 ml per hand injected by a blunt tip microcannula (25G or 22G, preferably 22G), with fanning technique through a single entry point performing 5 passages and injecting 0,3 ml per passage.
  Day 0: Information and consent form provided. Clinical photography, Clinical assessment, Instrumental assessment, First treatment of Profhilo® (refer to study protocol).
  Day 30 (1 month after day 0): Clinical photography, Clinical assessment, Instrumental assessment, Second treatment of Profhilo® (refer to study protocol), Self-evaluation questionnaire.
  Day 120 (4 months after day 0): Clinical photography, Clinical assessment, Instrumental assessment, NO treatment, Self-evaluation questionnaire.
  Interventions: Device: Profhilo® Body

INTERVENTIONS:
Device: Profhilo® Body — Dosage form: Profhilo® Body (IBSA Farmaceutici Italia S.r.l.) is a resorbable medical device 3.25 ml non-pyrogenic pre-filled syringe, containing 3 ml of 3.2% hyaluronic acid for intradermal use (48 mg H-HA + 48 mg L-HA) dissolved in 3 ml of saline buffered sodium chloride.

SUMMARY:
People lose collagen all over the body, not just in the face; skin roughness and laxity of the dorsum of the hands can result from chrono and photo-aging. This skin roughness and laxity can range from very mild to severe; injection procedures can provide new tone and firmness to the skin of the hand dorsum. Dermal fillers are the most used non-permanent injectable materials available today to correct skin flaccidity and roughness on the dorsum of the hands. They give immediate aesthetic effect due to elastic gel matrix injected and impart longer term effects due to bio stimulation, promoting new collagen formation. The objective of this study is to investigate the aesthetic performance of the Hyaluronic acid (HA)- based dermal filler Profhilo® Body injected by a blunt tip microcannula (25G or 22G, preferably 22G), with fanning technique through a single entry point performing 5 passages and injecting 0,3 ml per passage, 1,5 ml for each hand. Volunteers of both sexes, aged 18-65 years with mild-moderate skin roughness and laxity at the level of hand dorsum are to be treated.

DETAILED DESCRIPTION:
Open, monocentric. 3 visits, 55 subjects.

Primary endpoint of the study is the evaluation of performance and tolerance of Profhilo Body (3ml) treatment in the back of the hands ( or dorsum of the hands). Secondary endpoint is self-assessment questionnaire by both doctors and volunteers.

Profhilo® Body (IBSA Farmaceutici Italia S.r.l.) is a resorbable medical device 3.25 ml non-pyrogenic pre-filled syringe, containing 3 ml of 3.2% hyaluronic acid for intradermal use (48 mg H-HA + 48 mg L-HA) dissolved in 3 ml of saline buffered sodium chloride. - IBSA Farmaceutici Italia S.r.l. - ITALY. The principle component is cross-linked Hyaluronic Acid of non-animal origin, produced by bacterial fermentation.

ELIGIBILITY:
Inclusion Criteria: Will be included in the study volunteers with the following characteristics:

* female and male sex, not necessarily 1:1 ratio;
* age 18-65 years;
* asking for hands restoration;
* available and able to return to the study site for the post-procedural follow-up examinations;
* accepting to not change their habits regarding food, physical activity, cosmetic and cleansing products for the hands;
* accepting not to expose their hands to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study, without appropriate sun protection;

Exclusion Criteria:

* Pregnancy;
* lactation;
* smokers;
* alcohol or drug abusers;
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* Body Mass Index (BMI) variation (± 1) during the study period;
* performing non-surgical skin aesthetic procedures for hands in the 6 months prior to the study start;
* aesthetic surgical procedure for the hands in the past;
* change in the normal habits regarding food, physical activity, cosmetic products and cleansing for the hands during the month preceding the test;
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit);
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study currently or during the previous 6 months.)
* presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* clinical and significant skin condition on the test area (e.g. active eczema, psoriasis, sclerodermia, local infections).

Exclusion criteria due to systemic disease:

* Diabetes;
* endocrine disease;
* hepatic disorder;
* renal disorder;
* cardiac disorder;
* pulmonary disease;
* cancer;
* neurological or psychological disease;
* inflammatory/immunosuppressive disease;
* drug allergy Exclusion criteria due to ongoing pharmacological treatment
* Anticoagulants and antiplatelet drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago);
* using of drugs able to influence the test results in the investigator opinion. The use of other drugs, not mentioned above, can be authorized by the Investigator. The trade name, the dosage, the start and stop date of the therapy will be reported on concomitant medication form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Skin Roughness and flaccidity at 30 days and at 120 days post-injection | Day 0, Day 30, Day 120
  Visual score from 1 (no roughness and flaccidity) to 5 (very severe roughness and flaccidity)
Change from Baseline of Skin density (profilometry) at 30 days and at 120 days post-injection | Day 0, Day 30, Day 120
  A picture of the skin is taken thanks to Primos compact portable device (GFMesstechnik) and a 3D representation is elaborated by Primos software.
Change from Baseline of Superficial and deep skin plastoelasticity at 30 days and at 120 days post-injection | Day 0, Day 30, Day 120
  Measurement of the principal torsiometric parameters Ue (immediate extensibility), Uf (final extensibility), Uv (viscoelasticity) and Ur (immediate elastic recovery) by the instrument Dermal Torque Meter (Dia-Stron Ltd., UK)
Change from Baseline of Tissue dielectric constant value of superficial and deep skin layers at 30 days and at 120 days post-injection | Day 0, Day 30, Day 120
  Non-invasive measurements of dielectric constant of the skin and subcutaneous fat by MoistureMeterD (Delfin Technologies, Kuopio - Finland). MoistureMeterD measures the changes in the total water content in the tissue with 0.5mm and 1.5mm probes.
Change from Baseline of Photographic evaluation at 30 days and at 120 days post-injection | Day 0, Day 30, Day 120
  2D pictures of the dorsum of both hands are taken in order to support the aesthetic result assessment

SECONDARY OUTCOMES:
Efficacy questionnaire | Day 30, Day 120
  Self-assessment questionnaire regarding skin roughness and laxity of the treated areas, skin suppleness, skin smoothness, skin hydration, skin lifting, contour redefinition/remodeling (score: very marked; marked; medium; light; absent)
Treatment tolerance questionnaire | Day 30, Day 120
  Self-assessment score: bad; poor; good; excellent

CONTACTS AND LOCATIONS:
Overall Officials: Adele Sparavigna, MD, Principal Investigator — DERMING S.r.l., Clinical Research and Bioengineering Institute
Locations (1):
- DERMING S.r.l., Clinical Research and Bioengineering Institute, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT05590364/Prot_SAP_000.pdf